CLINICAL TRIAL: NCT02309073
Title: PC Protocol: Preconceptional Screening Part 2
Brief Title: PC Protocol: Preconceptional Screening
Acronym: PC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, Professor, UMC Utrecht
Other Study IDs: 13-109
Record Dates: First submitted 2013-11-06; First posted 2014-12-05 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood will be drawn for later determination of various parameters. DNA will also be extracted.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- women with a regular indication for ART: In the present proposal we are aiming to include all normo-ovulatory women with a regular indication for ART.
- women undergoing donor insemination treatment: potential normal fertile control group

SUMMARY:
Background: Despite considerable progress in the field of assisted reproductive technology (ART) maximum pregnancy rates generally do not exceed 30%. Furthermore, substantial differences in pregnancy rates are seen between women starting ART from seemingly similar clinical starting points and information on pregnancy/neonatal complications after ART is limited. For physicians and patients it would be extremely valuable if tools could be developed through which individualised chances of live birth and the development of pregnancy/neonatal complications can be calculated. In addition, there is increasing knowledge about health risks associated with subfertility and in particular with polycystic ovarian syndrome (PCOS) and premature ovarian failure (POF). An important void in research to date is the absence of a control group to check important new findings.

Objectives: The study protocol aims to form a cohort of normo-ovulatory women with a regular indication for ART which can aid the investigators principle lines of research:

1. To study initial predictors of ovarian response to stimulation for IVF
2. To study predictors of chances for live birth after repeated IVF cycles
3. To assess the role for vascular health in the probabilities of success in ART treatment
4. To study predictors for pregnancy and neonatal complications
5. To form a control group for cycle disturbance studies

Study design: In this part of the protocol, serum and material for DNA analysis will be collected by asking patients to have 20 ml of blood drawn during a routine blood withdrawal. This blood will be stored in the Biobank of the UMC Utrecht at -80 C.

Study population: All women starting ART will be asked to participate. Women starting donorinsemination treatment will be asked to participate, from the viewpoint that they potentially will form a normal fertile control group.

Nature and extent of the burden and benefits associated with participation: There are no benefits or risks for the study patient as blood is withdrawn during a routine venapuncture and results will not be used for clinical practice.

DETAILED DESCRIPTION:
The aim of this protocol is to collect serum and genotype from normo-ovulatory women with a regular indication for IVF/ICSI that can aid further research into the investigators principle lines of research which include improving performance ART treatment , limiting pregnancy complications, and improving offspring health.

ELIGIBILITY:
Inclusion Criteria:

* normo-ovulatory with a regular indication for ART or undergoing donorinsemination

Exclusion Criteria:

* Women with cycle disturbances

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the present proposal we are aiming to include all normo-ovulatory women with a regular indication for ART or undergoing donorinsemination
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2013-11; Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Ovarian response | 3 years
  number of oocytes, number of cycle cancellations, poor response, hyper response

SECONDARY OUTCOMES:
Prediction of pregnancy | 3 years
  prediction of clinical and ongoing pregnancy and live birth
Adverse pregnancy outcome | 3 years
  Number of patients with adverse pregnancy outcome including pregnancy induced hypertension,pre-eclampsia, HELLP syndrome, diabetes, premature birth, intrauterine growth restriction

CONTACTS AND LOCATIONS:
Overall Officials: Bart Fauser, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Hamdine O, Eijkemans MJC, Lentjes EGW, Torrance HL, Macklon NS, Fauser BCJM, Broekmans FJ. Antimullerian hormone: prediction of cumulative live birth in gonadotropin-releasing hormone antagonist treatment for in vitro fertilization. Fertil Steril. 2015 Oct;104(4):891-898.e2. doi: 10.1016/j.fertnstert.2015.06.030. Epub 2015 Jul 18. PMID 26196233
- [Derived] Hamdine O, Eijkemans MJ, Lentjes EW, Torrance HL, Macklon NS, Fauser BC, Broekmans FJ. Ovarian response prediction in GnRH antagonist treatment for IVF using anti-Mullerian hormone. Hum Reprod. 2015 Jan;30(1):170-8. doi: 10.1093/humrep/deu266. Epub 2014 Oct 29. PMID 25355590